CLINICAL TRIAL: NCT02032823
Title: A Randomised, Double-blind, Parallel Group, Placebo-controlled Multi-centre Phase III Study to Assess the Efficacy and Safety of Olaparib Versus Placebo as Adjuvant Treatment in Patients With gBRCA1/2 Mutations and High Risk HER2 Negative Primary Breast Cancer Who Have Completed Definitive Local Treatment and Neoadjuvant or Adjuvant Chemotherapy
Brief Title: Olaparib as Adjuvant Treatment in Patients With Germline BRCA Mutated High Risk HER2 Negative Primary Breast Cancer
Acronym: OlympiA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Breast International Group (Other); Frontier Science & Technology Research Foundation, Inc. (Industry); NRG Oncology (Other); Myriad Genetic Laboratories, Inc. (Industry); The Breast Adjuvant Study Team (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D081CC00006; NSABP B-55 (Other: NSABP); BIG 6-13 (Other: Breast International Group); 2024-511096-15-00 (Registry Identifier: Clinical Trail Information System (CTIS)); 2013-003839-30 (EudraCT Number)
Record Dates: First submitted 2014-01-03; First posted 2014-01-10 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Adjuvant; Olaparib; BRCA 1/2; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib (Experimental): Olaparib tablets 300mg b.i.d. p.o.
  Interventions: Drug: Olaparib
- Placebo (Placebo Comparator): Placebo tablets b.i.d. p.o.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olaparib — Patients will be administred olaparib orally twice daily (b.i.d.) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 ml of water
  Other Names: Lynparza
  Arms: Olaparib
Drug: Placebo — Patients will be administred matching placebo. Two (2) tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 ml of water
  Arms: Placebo

SUMMARY:
Olaparib treatment in patients with germline BRCA1/2 mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

DETAILED DESCRIPTION:
Patients will be randomised in 1:1 ratio to either olaparib or placebo. Randomisation will be stratified by Hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC), prior neoadjuvant versus adjuvant chemotherapy and prior platinum use for breast cancer.

Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months and 3 monthly for the remaining 6 months of study treatment plus 30 days after its discontinuation. Following randomisation, all patients will be assessed regularly for signs, symptoms and evidence of disease recurrence by taking medical history, physical examination and mammogram/breast MRI. Efficacy assessments will be performed on a 3 monthly basis during the first 2 years, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. All patients (except those with bilateral mastectomy) will have mammogram / breast MRI annually for 10 years beginning 6 months after randomisation.

All randomised patients will have clinical assessment visits for 10 years following their randomisation into the study. Once a patient completes 10 years of clinical assessment they will enter the survival follow up phase of the trial which will continue until approximately 10 years after the last patient is randomised.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast that is one of the following phenotypes:

  1. Triple negative breast cancer defined as: ER and PgR negative AND HER2 negative (not eligible for anti-HER2 therapy)
  2. ER and/or PgR positive, HER2 negative
* Documented germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
* Completed adequate breast and axilla surgery.
* Completed at least 6 cycles neoadjuvant or adjuvant chemotherapy containing anthracyclines, taxanes or the combination of both. Prior platinum as potentially curative treatment for prior cancer (e.g. ovarian) or as adjuvant or neoadjuvant treatment for breast cancer is allowed.
* ECOG 0-1.

Exclusion criteria:

* Any previous treatment with a PARP inhibitor, including olaparib and/or known hypersensitivity to any of the excipients of study treatment.
* Patients with second primary malignancy. EXCEPTIONS are:

  1. adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, Ductal Carcinoma in situ (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma
  2. other solid tumours and lymphomas (without bone marrow involvement) diagnosed ≥ 5 years prior to randomisation and treated with no evidence of disease recurrence and for whom no more than one line of chemotherapy was applied.
* Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Evidence of metastatic breast cancer

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1836 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2029-05-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tutt, Doctor of Medicine, Principal Investigator — Integrated Cancer Centre Guy's Hospital, King's College, London School of Medicine, London, UK; Judy Garber, Doctor of Medicine, Principal Investigator — Harvard Medical School, Center for Cancer Genetics and Prevention, Dana-Farber Cancer Institute, Susan F. Smither Center for Women's Cancers, 450 Brookline Avenue, Boston; MA 02215, US; Charles Geyer, Doctor of Medicine, Principal Investigator — Virginia Commonwealth University Massey Cancer Center, McGlothlin Medical Education Center, Room 12-217, 1201 East Marshall St., PO Box 980070, Richmond, VA 23298-0070, USA
Locations (601):
- United States (324):
  - Research Site, Anchorage, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Gilbert, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Baldwin Park, California
  - Research Site, Berkeley, California
  - Research Site, Duarte, California
  - Research Site, Fontana, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Los Angeles, California
  - Research Site, Martinez, California
  - Research Site, Newport Beach, California
  - Research Site, Oakland, California
  - Research Site, Palo Alto, California
  - Research Site, Paradise, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, San Jose, California
  - Research Site, San Leandro, California
  - Research Site, San Marcos, California
  - Research Site, Santa Cruz, California
  - Research Site, Santa Rosa, California
  - Research Site, South San Francisco, California
  - Research Site, Stockton, California
  - Research Site, Sunnyvale, California
  - Research Site, Vacaville, California
  - Research Site, Vallejo, California
  - Research Site, Woodland Hills, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Edwards, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Lafayette, Colorado
  - Research Site, Lone Tree, Colorado
  - Research Site, Derby, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Guilford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, North Haven, Connecticut
  - Research Site, Orange, Connecticut
  - Research Site, Torrington, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Daytona Beach, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Valdosta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Kuakini, Hawaii
  - Research Site, ‘Aiea, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Fruitland, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Nampa, Idaho
  - Research Site, Post Falls, Idaho
  - Research Site, Twin Falls, Idaho
  - Research Site, Centralia, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Effingham, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Glenview, Illinois
  - Research Site, Highland Park, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Mount Vernon, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Warrenville, Illinois
  - Research Site, Elkhart, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Mishawaka, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Plymouth, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Westville, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Bettendorf, Iowa
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Davenport, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Mason City, Iowa
  - Research Site, Chanute, Kansas
  - Research Site, El Dorado, Kansas
  - Research Site, Fairway, Kansas
  - Research Site, Garden City, Kansas
  - Research Site, Hays, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Lawrence, Kansas
  - Research Site, Newton, Kansas
  - Research Site, Olathe, Kansas
  - Research Site, Salina, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Winfield, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Houma, Louisiana
  - Research Site, Kenner, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Augusta, Maine
  - Research Site, Bangor, Maine
  - Research Site, Belfast, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Portland, Maine
  - Research Site, Rockport, Maine
  - Research Site, Sanford, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Easton, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Warren, Michigan
  - Research Site, Bemidji, Minnesota
  - Research Site, Burnsville, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Mankato, Minnesota
  - Research Site, Maple Grove, Minnesota
  - Research Site, Maplewood, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Shakopee, Minnesota
  - Research Site, Waconia, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Cape Girardeau, Missouri
  - Research Site, Joplin, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lee's Summit, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Norfolk, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Lebanon, New Hampshire
  - Research Site, Manchester, New Hampshire
  - Research Site, Nashua, New Hampshire
  - Research Site, Flemington, New Jersey
  - Research Site, Hamilton, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Mount Holly, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Charlotte, New York
  - Research Site, East Syracuse, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Albemarle, North Carolina
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Clinton, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Wilson, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Grand Forks, North Dakota
  - Research Site, Minot, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Beachwood, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Englewood, Ohio
  - Research Site, Findlay, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Oregon, Ohio
  - Research Site, Parma, Ohio
  - Research Site, Perrysburg, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Broomall, Pennsylvania
  - Research Site, Bryn Mawr, Pennsylvania
  - Research Site, Clairton, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Drexel Hill, Pennsylvania
  - Research Site, Ephrata, Pennsylvania
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Hazleton, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Lebanon, Pennsylvania
  - Research Site, Lewisburg, Pennsylvania
  - Research Site, Media, Pennsylvania
  - Research Site, Paoli, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, State College, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, Williamsport, Pennsylvania
  - Research Site, Wynnewood, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greenwood, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Temple, Texas
  - Research Site, American Fork, Utah
  - Research Site, Murray, Utah
  - Research Site, Ogden, Utah
  - Research Site, Provo, Utah
  - Research Site, St. George, Utah
  - Research Site, Berlin Corners, Vermont
  - Research Site, Burlington, Vermont
  - Research Site, Annandale, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Mechanicsville, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, South Hill, Virginia
  - Research Site, Centralia, Washington
  - Research Site, Kennewick, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Poulsbo, Washington
  - Research Site, Seattle, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Parkersburg, West Virginia
  - Research Site, Burlington, Wisconsin
  - Research Site, Chippewa Falls, Wisconsin
  - Research Site, Eau Claire, Wisconsin
  - Research Site, Elkhorn, Wisconsin
  - Research Site, Fond du Lac, Wisconsin
  - Research Site, Grafton, Wisconsin
  - Research Site, Green Bay, Wisconsin
  - Research Site, Kenosha, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Ladysmith, Wisconsin
  - Research Site, Marinette, Wisconsin
  - Research Site, Marshfield, Wisconsin
  - Research Site, Menomonee Falls, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Minocqua, Wisconsin
  - Research Site, Mukwonago, Wisconsin
  - Research Site, Oconomowoc, Wisconsin
  - Research Site, Rice Lake, Wisconsin
  - Research Site, Stevens Point, Wisconsin
  - Research Site, Summit, Wisconsin
  - Research Site, Waukesha, Wisconsin
  - Research Site, Wausau, Wisconsin
  - Research Site, Wauwatosa, Wisconsin
  - Research Site, West Allis, Wisconsin
  - Research Site, Weston, Wisconsin
  - Research Site, Wisconsin Rapids, Wisconsin
- Argentina (8):
  - Research Site, Berazategui
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, La Rioja
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (15):
  - Research Site, Adelaide
  - Research Site, Auchenflower
  - Research Site, Concord
  - Research Site, Douglas
  - Research Site, Gosford
  - Research Site, Hobart
  - Research Site, Malvern
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Randwick
  - Research Site, South Brisbane
  - Research Site, Tamworth
  - Research Site, Tweed Heads
  - Research Site, Waratah
  - Research Site, Wendouree
- Austria (13):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Rankweil
  - Research Site, Ried
  - Research Site, Salzburg
  - Research Site, Sankt Veit an der Glan
  - Research Site, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Weiz
  - Research Site, Wels
- Belgium (9):
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ostend
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- China (12):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
- France (23):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dechy
  - Research Site, La Roche-sur-Yon
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Plerin SUR MER
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Cloud
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (55):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Baden-Baden
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Bottrop
  - Research Site, Brandenburg
  - Research Site, Bremen
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Deggendorf
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Ebersberg
  - Research Site, Eggenfelden
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Fulda
  - Research Site, Fürth
  - Research Site, Gera
  - Research Site, Gifhorn
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hamelin
  - Research Site, Hanover
  - Research Site, Hildesheim
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Koblenz Am Rhein
  - Research Site, Leipzig
  - Research Site, Mainz Am Rhein
  - Research Site, Mannheim
  - Research Site, Memmingen
  - Research Site, Mühlhausen
  - Research Site, Mühlheim An Der Ruhr
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nordhausen
  - Research Site, Offenbach
  - Research Site, Onkologisch Hämatologische Sch
  - Research Site, Paderborn
  - Research Site, Ravensburg
  - Research Site, Recklinghausen
  - Research Site, Rostock
  - Research Site, Rotenburg (Wümme)
  - Research Site, Saarbrücken
  - Research Site, Schweinfurt
  - Research Site, Stendal
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Witten
- Research Site, Budapest, Hungary
- Research Site, Reykjavik, Iceland
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (19):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Bolzano
  - Research Site, Castellanza Varese
  - Research Site, Lecce
  - Research Site, Legnago
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Nehrar
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Prato
  - Research Site, Rimini
  - Research Site, Saronno
  - Research Site, Varese
  - Research Site, Viterbo
- Japan (22):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Morioka
  - Research Site, Nagoya
  - Research Site, Nankoku-shi
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Shizuoka
  - Research Site, Suita
- Netherlands (7):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Geleen
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Rotterdam
  - Research Site, Zaandam
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Grzepnica
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
- Research Site, San Juan, Puerto Rico
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (30):
  - Research Site, A Coruña
  - Research Site, Ávila
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Cáceres
  - Research Site, Córdoba
  - Research Site, Elche(Alicante)
  - Research Site, Girona
  - Research Site, Hosp de Llobregat(Barcelona)
  - Research Site, Jaén
  - Research Site, La Laguna (Tenerife)
  - Research Site, Lleida
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Reus,Tarragona
  - Research Site, Sabadell(Barcelona)
  - Research Site, Salamanca
  - Research Site, San Sebastián
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Terrassa(Barcelona)
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Malmo
  - Research Site, Solna
  - Research Site, Stockholm
  - Research Site, Umeå
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Zurich
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (18):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Dudley
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Southampton
  - Research Site, Stoke-on-Trent
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ganz PA, Bandos H, Spanic T, Friedman S, Muller V, Kuemmel S, Delaloge S, Brain E, Toi M, Yamauchi H, de Duenas EM, Armstrong A, Im SA, Song CG, Zheng H, Sarosiek T, Sharma P, Geng C, Fu P, Rhiem K, Frauchiger-Heuer H, Wimberger P, t'Kint de Roodenbeke D, Liao N, Goodwin A, Chakiba-Brugere C, Friedlander M, Lee KS, Giacchetti S, Takano T, Henao-Carrasco F, Virani S, Valdes-Albini F, Domchek SM, Bane C, McCarron EC, Mita M, Rossi G, Rastogi P, Fielding A, Gelber RD, Scheepers ED, Cameron D, Garber J, Geyer CE, Tutt ANJ. Patient-Reported Outcomes in OlympiA: A Phase III, Randomized, Placebo-Controlled Trial of Adjuvant Olaparib in gBRCA1/2 Mutations and High-Risk Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer. J Clin Oncol. 2024 Apr 10;42(11):1288-1300. doi: 10.1200/JCO.23.01214. Epub 2024 Feb 1. PMID 38301187
- [Derived] Perachino M, Poggio F, Arecco L, Blondeaux E, Spinaci S, Marrocco C, Levaggi A, Lambertini M. Update on Pregnancy Following Breast Cancer Diagnosis and Treatment. Cancer J. 2022 May-Jun 01;28(3):176-182. doi: 10.1097/PPO.0000000000000599. PMID 35594464
- [Derived] Tutt ANJ, Garber JE, Kaufman B, Viale G, Fumagalli D, Rastogi P, Gelber RD, de Azambuja E, Fielding A, Balmana J, Domchek SM, Gelmon KA, Hollingsworth SJ, Korde LA, Linderholm B, Bandos H, Senkus E, Suga JM, Shao Z, Pippas AW, Nowecki Z, Huzarski T, Ganz PA, Lucas PC, Baker N, Loibl S, McConnell R, Piccart M, Schmutzler R, Steger GG, Costantino JP, Arahmani A, Wolmark N, McFadden E, Karantza V, Lakhani SR, Yothers G, Campbell C, Geyer CE Jr; OlympiA Clinical Trial Steering Committee and Investigators. Adjuvant Olaparib for Patients with BRCA1- or BRCA2-Mutated Breast Cancer. N Engl J Med. 2021 Jun 24;384(25):2394-2405. doi: 10.1056/NEJMoa2105215. Epub 2021 Jun 3. PMID 34081848
- See also: AstraZeneca Cancer Study Locator Service Phone: 877 400 4656 Email: astrazeneca@emergingmed.com — http://www.emergingmed.com/networks/AstraZeneca
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081CC00006&attachmentIdentifier=dee7be50-99d3-44f3-8f8a-ffb3ca728507&fileName=Olympia_CTT_Redacted_Protocols_and_SAP_23Sept2021_PDF_A_Redacted_final.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 22 April 2014. Patients were randomised from 554 centres in 23 countries worldwide.
Pre-assignment Details: Patients with unknown germline BRCA (gBRCA) mutation status prior to randomisation underwent Screening Part 1 to ascertain gBRCA mutation status during, or prior to, neoadjuvant/adjuvant chemotherapy. All patients with known gBRCA mutation status (including those found through Screening Part 1) underwent Screening Part 2.
Groups:
- Olaparib: Olaparib tablets 300mg taken orally twice daily.
- Placebo: Placebo tablets taken orally twice daily.
Period: Overall Study
Arm/Group | Olaparib | Placebo
Started | 921 | 915
Completed | 0 | 0
Not Completed | 921 | 915
Not completed — Death | 75 | 109
Not completed — Lost to Follow-up | 18 | 17
Not completed — Withdrawal by Subject | 70 | 53
Not completed — Ongoing study at data cut-off | 755 | 731
Not completed — Other (e.g investigators decision, protocol deviation, randomised by mistake) | 3 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib | Placebo | Total
Number analyzed (Participants) | 921 | 915 | 1836
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (9.8) | 43.6 (10.1) | 43.3 (10.0)
Age, Customized [Number; unit: Participants]
  <30 years | 51 | 59 | 110
  30-39 years | 333 | 306 | 639
  40-49 years | 315 | 308 | 623
  50-59 years | 166 | 172 | 338
  60-69 years | 48 | 66 | 114
  >=70 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 919 | 911 | 1830
  Male | 2 | 4 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 34 | 24 | 58
  NOT HISPANIC OR LATINO | 805 | 812 | 1617
  NOT KNOWN, NOT RECORDED, OR REFUSED | 82 | 79 | 161
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 3 | 1 | 4
  ASIAN | 259 | 272 | 531
  BLACK OR AFRICAN AMERICAN | 19 | 29 | 48
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 1
  WHITE | 626 | 599 | 1225
  OTHER | 3 | 6 | 9
  MISSING | 10 | 8 | 18
Region of Enrollment [Number; unit: Participants]
  Argentina | 16 | 12 | 28
  Australia | 30 | 30 | 60
  Austria | 28 | 25 | 53
  Belgium | 12 | 26 | 38
  Canada | 11 | 23 | 34
  China | 117 | 130 | 247
  France | 77 | 65 | 142
  Germany | 106 | 92 | 198
  United Kingdom | 60 | 46 | 106
  Hungary | 8 | 9 | 17
  Iceland | 5 | 1 | 6
  Israel | 30 | 35 | 65
  Italy | 30 | 27 | 57
  Japan | 64 | 76 | 140
  Netherlands | 11 | 18 | 29
  Poland | 50 | 59 | 109
  Portugal | 7 | 6 | 13
  Korea, Republic Of | 53 | 44 | 97
  Spain | 63 | 46 | 109
  Sweden | 20 | 15 | 35
  Switzerland | 4 | 17 | 21
  Taiwan, Province Of China | 8 | 4 | 12
  United States | 111 | 109 | 220

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease Free Survival (IDFS)
Description: An IDFS event is defined as the first occurrence of loco-regional or distant recurrence or new cancer or death from any cause.
Time Frame: From date of randomisation to data cut off: 27 March 2020 (approximately 5 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 921 | 915
Participants | 106 | 178
Statistical Analysis 1: Comparison: Olaparib vs Placebo; Test type: Superiority; p = 0.0000073, Log Rank — A multiple testing procedure is employed across the primary and all key secondary endpoints to strongly control overall type I error at 5% (2 sided) accounting for all analysis timepoints; Log rank test is stratified by chemotherapy type, hormone receptor status, and prior platinum therapy using a pre-specified pooling strategy; Hazard Ratio (HR) = 0.581, 99.5% CI 2-sided [0.409 to 0.816] — Estimate of the treatment hazard ratio is based on a stratified Cox's Proportional Hazards Model, <1 indicates a lower risk with olaparib compared with placebo arm. Stratification factors are the same as those used in the stratified log-rank test

2. Secondary Outcome: Distant Disease Free Survival (DDFS)
Description: A DDFS event is defined as documented evidence of first distant recurrence of breast cancer or death from any cause
Time Frame: From date of randomisation to data cut off: 27 March 2020 (approximately 5 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 921 | 915
Participants | 89 | 152
Statistical Analysis 1: Comparison: Olaparib vs Placebo; Test type: Superiority; p = 0.0000257, Log Rank — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.574, 99.5% CI 2-sided [0.392 to 0.831] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival (OS)
Description: An OS event is defined as death by any cause.
Time Frame: From date of randomisation to data cut off: 12 July 2021 (approximately 7 years 3 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 921 | 915
Participants | 75 | 109
Statistical Analysis 1: Comparison: Olaparib vs Placebo; Test type: Superiority; p = 0.0091, Log Rank — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.678, 98.5% CI 2-sided [0.468 to 0.973] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Contralateral Invasive and Non-invasive Breast Cancer, New Primary Ovarian Cancer, New Primary Fallopian Tube Cancer and New Primary Peritoneal Cancer
Description: Number of patients with contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer. Analysis of contralateral breast cancers exclude patients with a bilateral mastectomy prior to randomisation. Analysis of new primary ovarian cancers excludes male patients and patients with a bilateral oophorectomy prior to randomisation. Analysis of new primary fallopian tube cancer excludes male patients and patients with a bilateral salpingectomy prior to randomisation. Analysis of new primary peritoneal cancers excludes male patients.
Time Frame: From date of randomisation to data cut off: 12 July 2021 (approximately 7 years 3 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 921 | 915
Participants
  Contralateral invasive breast cancer: number analyzed (Participants) | 583 | 597
  Contralateral invasive breast cancer | 19 | 21
  Contralateral non-invasive breast cancer: number analyzed (Participants) | 583 | 597
  Contralateral non-invasive breast cancer | 2 | 4
  New primary ovarian cancer: number analyzed (Participants) | 735 | 747
  New primary ovarian cancer | 1 | 5
  New primary fallopian tube cancer: number analyzed (Participants) | 756 | 758
  New primary fallopian tube cancer | 1 | 4
  New primary peritoneal cancer: number analyzed (Participants) | 919 | 911
  New primary peritoneal cancer | 0 | 0

5. Secondary Outcome: Change From Baseline for FACIT-Fatigue (Functional Assessment of Chronic Illness Therapy-Fatigue) Score for Participants Who Completed Neoadjuvant Chemotherapy
Description: Change from baseline for FACIT-Fatigue Score at 6, 12, 18 and 24 months for patients who completed neoadjuvant chemotherapy. Adjusted least-square mean changes and 95% Confidence Interval (CI) are obtained from mixed model for repeated measures (MMRM) analysis of the change from baseline. Only patients with evaluable baseline forms are included. FACIT-Fatigue score ranges from 0 to 52 with higher score indicating less fatigue.
Time Frame: 6, 12, 18 and 24 months after randomisation (data cut off: 12 July 2021)
Population: Patient reported outcomes (PRO) Analysis Set
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 382 | 359
Scores on a scale
  Change from baseline FACIT-Fatigue Score to 6 months | -1.5 [-2.3 to -0.8] | -0.2 [-1.0 to 0.6]
  Change from baseline FACIT-Fatigue Score to 12 months: number analyzed (Participants) | 382 | 356
  Change from baseline FACIT-Fatigue Score to 12 months | -1.5 [-2.4 to -0.6] | 0.0 [-0.9 to 0.9]
  Change from baseline FACIT-Fatigue Score to 18 months | 1.3 [0.4 to 2.2] | 1.4 [0.5 to 2.3]
  Change from baseline FACIT-Fatigue Score to 24 months | 1.6 [0.7 to 2.4] | 2.0 [1.1 to 2.9]

6. Secondary Outcome: Change From Baseline for FACIT-Fatigue (Functional Assessment of Chronic Illness Therapy-Fatigue) Score for Participants Who Completed Adjuvant Chemotherapy
Description: Change from baseline for FACIT-Fatigue Score at 6, 12, 18 and 24 months for patients who completed adjuvant chemotherapy. Adjusted least-square mean changes and 95% CI are obtained from mixed model for repeated measures (MMRM) analysis of the change from baseline. Only patients with evaluable baseline forms are included. FACIT-Fatigue score ranges from 0 to 52 with higher score indicating less fatigue.
Time Frame: 6, 12, 18 and 24 months after randomisation (data cut off: 12 July 2021)
Population: Patient reported outcomes (PRO) Analysis Set
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 382 | 406
Scores on a scale
  Change from baseline FACIT-Fatigue Score to 6 months | -0.7 [-1.5 to 0.0] | 0.6 [-0.2 to 1.3]
  Change from baseline FACIT-Fatigue Score to 12 months | -0.8 [-1.6 to 0.0] | 0.5 [-0.3 to 1.2]
  Change from baseline FACIT-Fatigue Score to 18 months | 0.9 [0.1 to 1.7] | 1.2 [0.4 to 2.0]
  Change from baseline FACIT-Fatigue Score to 24 months | 1.3 [0.5 to 2.1] | 1.6 [0.7 to 2.4]

7. Secondary Outcome: Change From Baseline for EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core Questions 30) Scores for Participants Who Completed Neoadjuvant Chemotherapy
Description: Change from baseline for EORTC QLQ-C30 Global health status QOL (Quality of Life) Score at 6, 12, 18 and 24 months for patients who completed neoadjuvant chemotherapy. Adjusted least-square mean changes and 95% CI are obtained from mixed model for repeated measures (MMRM) analysis of the change from baseline. Only patients with evaluable baseline forms are included. EORTC QLQ-C30 scores range from 0 to 100 with higher score indicating better quality of life.
Time Frame: 6, 12, 18 and 24 months after randomisation (data cut off: 12 July 2021)
Population: Patient reported outcomes (PRO) Analysis Set
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 382 | 358
Scores on a scale
  Change from baseline EORTC QLQ-C30 Global health status score to 6 months | -0.4 [-2.2 to 1.4] | 0.4 [-1.4 to 2.2]
  Change from baseline EORTC QLQ-C30 Global health status score to 12 months | 0.5 [-1.5 to 2.4] | 2.7 [0.7 to 4.7]
  Change from baseline EORTC QLQ-C30 Global health status score to 18 months | 3.3 [1.3 to 5.3] | 4.4 [2.3 to 6.4]
  Change from baseline EORTC QLQ-C30 Global health status score to 24 months | 2.8 [0.6 to 5.0] | 6.1 [3.8 to 8.4]

8. Secondary Outcome: Change From Baseline for EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core Questions 30) Scores for Participants Who Completed Adjuvant Chemotherapy
Description: Change from baseline for EORTC QLQ-C30 Global health status QOL (Quality of Life) Score at 6, 12, 18 and 24 months for patients who completed adjuvant chemotherapy. Adjusted least-square mean changes and 95% CI are obtained from mixed model for repeated measures (MMRM) analysis of the change from baseline. Only patients with evaluable baseline forms are included. EORTC QLQ-C30 scores range from 0 to 100 with higher score indicating better quality of life.
Time Frame: 6, 12, 18 and 24 months after randomisation (data cut off: 12 July 2021)
Population: Patient reported outcomes (PRO) Analysis Set
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olaparib | Placebo
Number analyzed (Participants) | 383 | 407
Scores on a scale
  Change from baseline EORTC QLQ-C30 Global health status score to 6 months | -0.5 [-2.2 to 1.2] | 2.2 [0.6 to 3.8]
  Change from baseline EORTC QLQ-C30 Global health status score to 12 months | 0.6 [-1.1 to 2.4] | 3.1 [1.5 to 4.8]
  Change from baseline EORTC QLQ-C30 Global health status score to 18 months | 2.9 [1.1 to 4.7] | 5.1 [3.3 to 6.9]
  Change from baseline EORTC QLQ-C30 Global health status score to 24 months | 4.5 [2.6 to 6.4] | 4.8 [2.9 to 6.7]

ADVERSE EVENTS:
Time Frame: Maximum of approximately 13 months.
Description: All-Cause Mortality was collected for the Full Analysis Set (FAS). Serious and Other Adverse Events were collected for the Safety Analysis Set (SAS), which includes all participants who received at least 1 dose of randomized study treatment (N=1815). There were 10 patients in the olaparib arm and 11 patients in the placebo arm that did not receive study treatment and therefore are excluded from the SAS. The Other Adverse Events section reports AE's of any grade where the frequency is above 5%.
Groups:
- Olaparib; Placebo: Description (Arm-group)
Arm/Group | Olaparib | Placebo
All-Cause Mortality (participants affected / at risk) | 75/921 | 109/915
Serious Adverse Events (participants affected / at risk) | 79/911 | 78/904
Other Adverse Events (participants affected / at risk) | 793/911 | 672/904
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib (N=911) | Placebo (N=904)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Vith nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 15 (17) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (5) | 0 (0)
Foreign body reaction (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 3 (3) | 6 (6)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Fallopian tube cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib (N=911) | Placebo (N=904)
Insomnia (Psychiatric disorders) | 67 (71) | 61 (65)
Cough (Respiratory, thoracic and mediastinal disorders) | 77 (85) | 72 (80)
Hot flush (Vascular disorders) | 73 (76) | 74 (76)
Abdominal pain (Gastrointestinal disorders) | 86 (96) | 65 (77)
Anaemia (Blood and lymphatic system disorders) | 201 (262) | 34 (39)
Constipation (Gastrointestinal disorders) | 84 (89) | 78 (88)
Diarrhoea (Gastrointestinal disorders) | 160 (198) | 124 (162)
Dyspepsia (Gastrointestinal disorders) | 55 (62) | 37 (39)
Nausea (Gastrointestinal disorders) | 519 (683) | 213 (267)
Stomatitis (Gastrointestinal disorders) | 81 (116) | 36 (38)
Vomiting (Gastrointestinal disorders) | 204 (294) | 74 (84)
Fatigue (General disorders) | 366 (442) | 248 (288)
Influenza like illness (General disorders) | 58 (65) | 44 (56)
Pain (General disorders) | 68 (78) | 74 (83)
Pyrexia (General disorders) | 48 (57) | 39 (44)
Nasopharyngitis (Infections and infestations) | 31 (45) | 52 (74)
Upper respiratory tract infection (Infections and infestations) | 79 (92) | 75 (104)
Lymphocyte count decreased (Investigations) | 62 (88) | 15 (16)
Neutrophil count decreased (Investigations) | 146 (211) | 59 (80)
White blood cell count decreased (Investigations) | 144 (213) | 52 (69)
Decreased appetite (Metabolism and nutrition disorders) | 119 (135) | 53 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 89 (95) | 115 (127)
Back pain (Musculoskeletal and connective tissue disorders) | 60 (65) | 72 (76)
Myalgia (Musculoskeletal and connective tissue disorders) | 50 (58) | 49 (50)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62 (74) | 64 (70)
Dizziness (Nervous system disorders) | 104 (113) | 66 (72)
Dysgeusia (Nervous system disorders) | 107 (125) | 38 (41)
Headache (Nervous system disorders) | 178 (217) | 151 (195)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions are imposed by the trial's Steering Committee (SC) and intend to ensure that all publications/presentations are peer reviewed by the SC. Sponsor has the right to review/comment on the content of the material to be published/presented, may request removal of confidential information (e.g. patentable information/trade secrets) within max 90 days. Individual Institutions may publish/present data from their site(s) in compliance with conditions defined in Study Publication Policy.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT02032823/Prot_SAP_000.pdf